CLINICAL TRIAL: NCT05365646
Title: Fall Risk Assessment and Speech Intelligibility Enhancement Using In-ear Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Starkey Laboratories, Inc (Industry)
Responsible Party: Principal Investigator, Kristen K. Steenerson, MD, Clinical Associate Professor in Otoneurology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 60900
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss; Dizziness; Vertigo; Fall Related Injury Risk; Fall Prevention; Imbalance; Speech Intelligibility
Keywords: Fall risk; Hearing loss
MeSH Terms: conditions — Hearing Loss; Dizziness; Vertigo; Speech Intelligibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Fall risk assessment (Experimental): Participants will wear study hearing aids that are equipped with embedded sensors and artificial intelligence. This will help track their movement and signal if the participant falls or is at fall risk.
  Interventions: Device: Hearing aids equipped with motion sensing abilities
- Speech intelligibility (Experimental): Participants will wear study hearing aids that are equipped with embedded sensors and artificial intelligence. This will help track their movement and signal if the participant falls or is at fall risk.
  Interventions: Device: Hearing aids equipped with motion sensing abilities

INTERVENTIONS:
Device: Hearing aids equipped with motion sensing abilities — Participants will wear hearing aids that will assess their movement, and fall risk.

SUMMARY:
The purpose of this study is to develop and validate methods to use hearing aids equipped with embedded sensors and artificial intelligence to assist in the assessment of fall risk and in the implementation of interventions aimed at reducing the risk of falling, as well as to improve speech intelligibility in quiet and in background noise, track physical activity, and social engagement. The investigators hope is that the knowledge that is generated through this study will ultimately translate to the clinical setting and will help reduce the likelihood that individuals experience a fall, and improve the quality of hearing in individuals who wear hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Bilateral hearing aid user
* Able to consent in English
* Having access to a phone capable of running the mobile app required for the study
* Screen for fall risk ("Yes" to any question: Feels unsteady when standing or walking? Worries about falling? Has fallen in past year? If the participant has fallen: how many times? were they injured/hurt?)
* Ambulatory without need for a wheelchair

Exclusion Criteria:

* People with mobility restrictions (e.g., wheelchair bound) that would prevent the performance of the functional assessments.
* People with severe movement (e.g., Advanced Parkinson's disease) or cognitive (e.g., advanced dementia) disorders that would prevent the individual from either performing the functional assessments, or would lead to restricted activities that would prevent motion data from being collected according to the goal of the study.
* Inability to understand, consent, and complete requirements including verbal instructions and non-ambulatory/wheelchair-dependent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fall risk assessment using CDC's STEADI protocol | approximately 15 minutes to assess
  Participants will undergo the Centers for Disease Control and Prevention (CDC)'s STEADI (Stopping Elderly Accidents, Deaths & Injuries) fall risk assessment with the hearing aids on. The scoring for these tests will be done by the tester, 2 independent raters, and the hearing aids. A comparison of the fall risk assessments by the testers and the hearing aids is the primary outcome measure. This outcome is assessed in Fall Risk Assessment participants only.
Timed Up and Go Test | approximately 15 minutes to assess
  Duration of time to stand, walk to a line on the floor (3 meters/10 feet away), turn around, return to chair and sit. Participants wear their regular footwear and can use a walking aid if needed. This outcome is assessed in Fall Risk Assessment participants only.
30-Second Chair Stand Test | approximately 15 minutes to assess
  Number of times participants can stand without using their arms during the test. Participants wear their regular footwear and can use a walking aid if needed. This outcome is assessed in Fall Risk Assessment participants only.
4-Stage Balance Test | approximately 15 minutes to assess
  Participants who are able to keep their balance for 10 second in each of four positions (feet together, feet staggered, feet in tandem, and single foot stand). They can hold their arms out, or move their body to help keep your balance, but not move their feet. This outcome is assessed in Fall Risk Assessment participants only.
Consonant-Nucleus-Consonant (CNC) | Approximately 10-15 minutes.
  The number and percentage of words and phonemes accurately repeated are measured in aided (using hearing aids) and unaided conditions. This outcome is measured in Speech Intelligibility participants only.
Quick Speech-in-Noise (QuickSIN) | Approximately 10-15 minutes.
  The number and percentage of words and phonemes accurately repeated are measured in ambient noise conditions in aided and unaided conditions. This outcome is measured in Speech Intelligibility participants only.
Words-in-Noise (WIN) | Approximately 10-15 minutes.
  The number and percentage of words and phonemes accurately repeated are measured in muli-talker babble noise conditions in aided and unaided conditions. This outcome is measured in Speech Intelligibility participants only.
Nonsense Syllable Test (NST) | Approximately 10-15 minutes.
  The number and percentage of words and phonemes accurately repeated are measured in continuous noise conditions in aided and unaided conditions. This outcome is measured in Speech Intelligibility participants only.

SECONDARY OUTCOMES:
Fall screening questionnaire using CDC's STEADI protocol | Approximately 2 minutes.
  Participants are screened using the CDC's "Three Key Questions" which are part of the STEADI Protocol.
Listening Effort Questionnaire Scale Score | Approximately 5 minutes.
  Listening effort scale score measures the participant's perceived listening effort. This outcome is measured in Speech Intelligibility participants only.
Auditory Lifestyle and Demand Scale Score | Approximately 5 minutes.
  Auditory Lifestyle and Demand scale score measures perceived demands of hearing on lifestyle. This outcome is measured in Speech Intelligibility participants only.
User Experience Questionnaire | Approximately 2 minutes.
  Participants rate their experience with the hearing aid regarding the following aspects: perceived difficulty communicating and listening effort in different environments.
Demographic and Health Questionnaires | Approximately 15 minutes.
  Data is gathered on age, sex, education level, hand-laterality, professional background, exercise habits, race, ethnicity, marital status, health literacy scores, medical conditions, and medications.
Orthostatic Blood Pressure | Approximately 15 minutes.
  Blood pressure measurements in laying down, sitting, and standing positions.
Pure-Tone Audiometry | Approximately 15 minutes.
  Hearing thresholds are measured from 250Hz through 8kHz in both ears, air and bone conduction.
Activities-Specific Balance Confidence Questionnaire | Approximately 10 minutes.
  Participants rate their confidence level in various balance situations.
Speech, Spatial Qualities of Hearing Scale (SSQ) | Approximately 10 minutes.
  Participants rate their difficulty level with understanding speech in various hearing situations.
Hearing Aid Data | Approximately 5 minutes.
  Data is gathered from the participants' hearing aids on wear-time, streaming time, time spent in various sound classes and software updates. Data is also collected on the participants' required receiver length and coupling, as well as any specific fitting requirements they may have.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Ear Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahme M, Folkeard P, Scollie S. Evaluating the Accuracy of Step Tracking and Fall Detection in the Starkey Livio Artificial Intelligence Hearing Aids: A Pilot Study. Am J Audiol. 2021 Mar 10;30(1):182-189. doi: 10.1044/2020_AJA-20-00105. Epub 2020 Dec 7. PMID 33284647
- [Background] Burwinkel JR, Xu B, Crukley J. Preliminary Examination of the Accuracy of a Fall Detection Device Embedded into Hearing Instruments. J Am Acad Audiol. 2020 Jun;31(6):393-403. doi: 10.3766/jaaa.19056. Epub 2020 Aug 3. PMID 31914373